CLINICAL TRIAL: NCT06043154
Title: Discovering New Insights Into Anorexia Nervosa: Influence of MicrObial DysbiosiS (DIAMOnDS)
Acronym: DIAMOnDS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Fondation de France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RC21_0598
Record Dates: First submitted 2023-09-04; First posted 2023-09-21 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Anorexia Nervosa
Keywords: microbiota, dysbiosis
MeSH Terms: conditions — Anorexia Nervosa; Dysbiosis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anorexia nervosa (Experimental)
  Interventions: Other: Patients with severe to extreme anorexia nervosa admitted to hospital for refeeding

INTERVENTIONS:
Other: Patients with severe to extreme anorexia nervosa admitted to hospital for refeeding — Clinical and biological measurements, blood and stool sample collection
  Other Names: Clinical and biological measurements, blood and stool sample collection

SUMMARY:
This study will investigate the link between the gut microbiota, the occurrence of the central adiposity phenotype, and the patients' fear to regain weight in anorexia nervosa.

DETAILED DESCRIPTION:
Excessive concerns about body shape and intense fear of becoming fat are among the core features of Anorexia Nervosa (AN). During refeeding, patients commonly report a disproportionate deposition of fat in the abdomen which could represent an obstacle for weight gain. It is not known whether these complaints are caused by dysmorphophobia or if the distribution of fat during refeeding could really not be uniform. Indeed, a "central adiposity phenotype" has already been objectified by anthropometric measures or imaging, with a higher proportion of visceral fat accumulated in the abdomen during the refeeding. This phenomenon could exacerbate body shape concerns and ultimately lead to an elevated risk of resistance to treatment and/or relapse.

The present research project aims to explore the mechanisms that underlie these difficulties, especially by investigating the link between the gut microbiota (both composition and products) and the occurrence of the central adiposity phenotype, and the patients' fear to regain weight.

Patients with severe to extreme anorexia nervosa admitted at hospital for refeeding will be included.

To describe patients included, a short clinical examination will be performed during the first week after inclusion, including several measures (sociodemographic data, medical history, history of eating disorders, current symptomatology of AN, and a dietary survey).

To investigate the gut microbiota biomarkers in stool (composition, diversity and richness, and metabolites), stool samples will be collected during the first week after inclusion and during the last week before discharge, together with information useful to stool sample analyses (related to stool consistency, intestinal transit, abdominal pain or discomfort, and psychoactive substance and prebiotics use).

In addition, blood samples will be collected during the first week after inclusion and during the last week before discharge, to investigate : (i) the levels of metabolites of the gut microbiota in blood, (ii) the nutritional and inflammation status.

To investigate central adiposity phenotype, anthropometric data will be collected weekly throughout the hospitalisation (including during the first and last week), and dual-energy X-ray absorptiometry (DXA) will be administered during the first week after inclusion and during the last week before discharge.

To investigate clinical outcomes, several self-reported questionnaires will be completed by the patients during the first week after inclusion and during the last week before discharge, including cognitive and behavioral characteristics of AN, body shape concerns, level of physical hyperactivity, anxiety and depression. Moreover, treatment-related data, hormonal situation and eating disorder episodes will be collected during weekly follow-up visits. Finally, a short clinical examination will be performed during the last week before discharge to collect the whole duration of hospitalisation and the current symptomatology of eating disorders.

This will allow to compare gut microbiota biomarkers (composition, diversity and richness, and metabolites) between patients with and without occurrence of the central adiposity phenotype during refeeding, to estimate the frequency of the occurrence of the central adiposity phenotype during refeeding, to characterise the gut microbiota biomarkers of patients with severe to extreme anorexia nervosa, to investigate the association between the occurrence of the central adiposity phenotype during the refeeding and clinical outcomes of the hospitalisation, to identify the gut microbiota biomarkers associated with clinical outcomes of the hospitalisation, and to estimate a mediation model to explain the links between the gut microbiota biomarkers and clinical outcomes, through the occurrence of the central adiposity phenotype and the change in body shape concerns..

An ancillary study will also be perfomed for patients participating to the DIAMOnDS study and accepting to participate to this ancillary study aimed at investigating the association between microbial and metabolic biomarkers of the gut microbiota (data collected in the DIAMOnDS study) and osteoporosis at inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Over 15 years old and 3 months.
* Admitted in the specialized department for eating disorders of CHU Nantes for refeeding.
* With a diagnosis of anorexia nervosa at admission (restrictive or Binge-Eating-Purging type).
* Body Mass Index at admission below 16 kilogram per square meter.
* Written informed consent for patients over 18 years old/ oral informed consent from both the patient and a legal representative for patients under 18 years old.
* Affiliated with French social security system or beneficiary from such system.

Exclusion Criteria:

* Pregnant and breastfeeding women.
* Who received a treatment with antibiotic/antifungal (other than local application) in the last three months.
* Who had a weight gain in the last month (5% or more of the patient's weight at admission).
* Under trusteeship or guardianship.
* Not fluent in French
* Who participate in another interventional study involving medication.
* Patients for whom stool collection or body mass composition analysis (with Dual-energy X-ray absorptiometry) couldn't be done during the first week of hospitalisation.

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Women only, due to the high influence of sex hormones and the low sex ratio of men admitted at hospital for anorexia nervosa.
Enrollment: 60 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Identification of gut microbiota biomarkers - composition | At inclusion
  Species-level taxonomic profile and functional potential of the gut microbiota generated by shotgun metagenomics performed on stool samples collected at inclusion, between those who express or not the central adiposity phenotype.
Identification of gut microbiota biomarkers - diversity and richness | At inclusion
  α-diversity, β-diversity, richness in genes, richness in species and enterotype of the gut microbiota generated by shotgun metagenomics performed on stool samples collected at inclusion, between those who express or not the central adiposity phenotype
Identification of gut microbiota biomarkers - metabolites | At inclusion
  Levels of Short Chain Fatty Acids (SCFAs) (acetate, propionate, butyrate, valerate, isobutyrate and isovalerate) produced by the gut microbiota estimated through gas chromatography-mass spectrometry on blood and stool samples collected at inclusion, between those who express or not the central adiposity phenotype.

SECONDARY OUTCOMES:
Identification of the central adiposity phenotype | At inclusion
  Proportion of patients who respond to the definition of the central adiposity phenotype during the refeeding. (The definition of the central adiposity phenotype will be characterised quantitatively through repeated measures of anthropometric data throughout the hospitalisation (waist-hip ratio (WHR), triceps skin fold, body mass index (BMI) and percentage from target weight) and qualitatively through Dual-energy X-ray Absorptiometry (DXA) imaging (repartition in body segment, relative proportion of lean and fat tissues, of subcutaneous and visceral fat mass, and of android and gynoid fat mass)).
Characterisation of gut microbiota biomarkers of patients with severe to extreme anorexia nervosa - composition | At inclusion
  species-level taxonomic profile and functional potential of the gut microbiota generated by shotgun metagenomics performed on stool samples collected at inclusion
Characterisation of gut microbiota biomarkers of patients with severe to extreme anorexia nervosa - diversity and richness | At inclusion
  α-diversity, β-diversity, richness in genes, richness in species and enterotype of the gut microbiota generated by shotgun metagenomics performed on stool samples collected at inclusion
Characterisation of gut microbiota biomarkers of patients with severe to extreme anorexia nervosa - metabolites | At inclusion
  levels of Short Chain Fatty Acids (SCFAs) (acetate, propionate, butyrate, valerate, isobutyrate and isovalerate) produced by the gut microbiota estimated through gas chromatography-mass spectrometry on blood and stool samples collected at inclusion
Variation of the composition of the gut microbiota between admission and discharge | At discharge, anticipated average 10 weeks
  Change in the species-level taxonomic profile and functional potential of the gut microbiota generated by shotgun metagenomics, between stool samples collected at inclusion and at discharge
Variation of the diversity and richness of the gut microbiota between admission and discharge | At discharge, anticipated average 10 weeks
  Change in the α-diversity, β-diversity, richness in genes, richness in species and enterotype of the gut microbiota generated by shotgun metagenomics, between stool samples collected at inclusion and at discharge
Variation of the metabolites of the gut microbiota between admission and discharge | At discharge, anticipated average 10 weeks
  Change in the levels of Short Chain Fatty Acids (SCFAs) (acetate, propionate, butyrate, valerate, isobutyrate and isovalerate) produced by the gut microbiota estimated through gas chromatography-mass spectrometry, between stool samples collected at inclusion and at discharge and between blood samples collected at inclusion and at discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: Undecided
undecided